CLINICAL TRIAL: NCT02759029
Title: Development of Treatment Algorithm for Eradication of Helicobacter Pylori Based on Antibiotic Susceptibility Test
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Jie hyun Kim, Associate Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3-2015-0193
Record Dates: First submitted 2016-04-26; First posted 2016-05-03 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-04

CONDITIONS: Helicobacter Pylori Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Susceptibility-guided group (Active Comparator): Drugs according to antimicrobial susceptibility-guided treatment
  Interventions: Drug: eradication of Helicobacter pylori
- triple therapy group (Sham Comparator): Drugs - Pantoloc 40mg, PO, BID, 1wk Amoxacillin 1g, PO, BID, 1wk Clarithromycin 500mg, PO, BID, 1wk
  Interventions: Drug: eradication of Helicobacter pylori
- concomitant therapy group (Sham Comparator): Drugs - Pantoloc 40mg, PO, BID, 1wk Amoxacillin 1g, PO, BID, 1wk Clarithromycin 500mg, PO, BID, 1wk Metronidazole 500mg, PO, BID, 1wk
  Interventions: Drug: eradication of Helicobacter pylori

INTERVENTIONS:
Drug: eradication of Helicobacter pylori — clarithromycin-based triple therapy Pantoloc 40mg, PO, BID, 1wk Amoxacillin 1g, PO, BID, 1wk Clarithromycin 500mg, PO, BID, 1wk
  * concomitant therapy group Pantoloc 40mg, PO, BID, 1wk Amoxacillin 1g, PO, BID, 1wk Clarithromycin 500mg, PO, BID, 1wk Metronidazole 500mg, PO, BID, 1wk
  * bismuth based quadraple therapy Pantoloc 40mg, PO, BID, 1wk Bismuth, 300mg, PO, QID, 1wk Tetracycline, 500mg, PO, QID, 1wk Metronidazole, 500mg, PO, TID, 1wk
  * levofloxacine based triple therapy Pantoloc 40mg, PO, BID, 1wk Amoxacillin 1g, PO, BID, 1wk Levofloxacin 500mg, PO, QD, 1wk

SUMMARY:
Helicobacter pylori eradication (H. pylori) rates with clarithromycin-based triple therapy are declining, and an alternative strategy is needed urgently. The investigators sought to compare the efficacy of pretreatment antimicrobial susceptibility-guided vs. clarithromycin-based triple therapy vs. concomitant therapy for H. pylori eradication in a region with high rates of multiple drug resistance.

ELIGIBILITY:
Inclusion Criteria:

1. positive results of rapid urease test

Exclusion Criteria:

1. liver cirrhosis,
2. chronic kidney disease,
3. bleeding tendency,
4. pregnant,
5. allergy to antibiotics

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
eradication rate of Helicobacter pylori | the H. pylori status was checked 4 weeks aft er the end of treatment using the 13 C-urea breath test.

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided